CLINICAL TRIAL: NCT04698993
Title: Dräger Antigen Test SARS-CoV-2 Clinical Performance Study
Brief Title: Dräger COVID-19 Antigen Test Clinical Performance Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: poor recruitment
Sponsor: Drägerwerk AG & Co. KGaA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Dräger Antigen Test SARS-CoV-2
Record Dates: First submitted 2021-01-05; First posted 2021-01-07 (Actual); Results first posted 2021-06-25 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Covid19
Keywords: antigen test
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Symptomatic (Other): Collection of specimens from symptomatic COVID-19 positive participants
  Interventions: Diagnostic Test: Dräger Antigen Test SARS-CoV-2
- Asymptomatic (Other): Collection of specimens from asymptomatic participants who had known or suspected exposure to SARS-CoV-2
  Interventions: Diagnostic Test: Dräger Antigen Test SARS-CoV-2

INTERVENTIONS:
Diagnostic Test: Dräger Antigen Test SARS-CoV-2 — Collection of patient samples using the Dräger sample collector with subsequent test reading via the Dräger Antigen SARS-CoV-2 Test

SUMMARY:
The study is designed to demonstrate suitability of the Dräger Antigen Test for SARS-CoV-2 detection in clinical nasal specimens. Real-time polymerase chain reaction (RT-PCR) on specimens collected by pharyngeal swabs serves as a reference method.

DETAILED DESCRIPTION:
The Dräger Antigen Test SARS-CoV-2 is a rapid lateral flow immunoassay for the qualitative detection of SARS-CoV-2 nucleoprotein directly from less invasive nasal swabs, to be performed at the point of care. The test kit contains all components required to carry out a test detecting SARS-CoV-2 nucleoprotein.

The study is designed to demonstrate suitability of the Dräger Antigen Test for SARS-CoV-2 detection in clinical nasal specimens. Real-time polymerase chain reaction (RT-PCR) on specimens collected by pharyngeal swabs serves as a reference method.

The goal of the study is to compare Dräger test results to the corresponding PCR data for overall sensitivity and specificity. Specimens are collected from patients showing COVID-19 symptoms as well as asymptomatic participants. Participants are recruited across all genders and eligible age groups. Study staff records participants' information such as symptoms and time since symptom onset. For each study participant, the specimen for RT-PCR is collected first, then the Dräger test specimen. The Dräger test result is read after 15 min to 20 min.

ELIGIBILITY:
Inclusion Criteria:

* Participants must require SARS-CoV-2 testing for the following reasons:

  * COVID-19 symptoms (Fever, cough and/or sore throat, fatigue/ general feeling of weakness, loss of sense of smell and/or taste, shortness of breath, muscle stiffness/ body aches, head cold/ running nose, etc.) on the day of testing, or
  * Known or suspected exposure to SARS-CoV-2 (contact persons etc.), or
  * Member of a group of high risk of exposure such as healthcare workers etc., or
  * Require screening for any other reason, e.g. doctor's orders, hygiene directive etc.
* Participant must be of legal age and must be able to understand the procedure and letter of consent.

Exclusion Criteria:

* Patients younger than 18 years old are excluded from the study.
* Pregnant or breastfeeding patients are excluded from the study.
* Patients unable to provide written informed consent are excluded.
* Patients with bleeding disorder are excluded from the study as a precaution.
* Hospitalized patients/inpatients are excluded.
* Application of nasal spray within 15 min prior to testing.
* Participants with symptoms on the day of testing are excluded, if any of their symptoms started more than 14 days prior to testing.
* Asymptomatic participants are excluded, if they experienced any symptoms in the 14 days prior to testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2021-03-22 (Actual); Study Completion 2021-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Zickler, Dr, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Symptomatic | Asymptomatic
Started | 275 | 113
Completed | 272 | 106
Not Completed | 3 | 7
Not completed — PCR results not accessible | 2 | 7
Not completed — incomplete documentation of kit assessment prior to testing | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Symptomatic | Asymptomatic | Total
Number analyzed (Participants) | 275 | 113 | 388
Age, Continuous [Mean (Full Range); unit: years] | 34.6 [18 to 73] | 32.5 [18 to 61] | 34.0 [18 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 66 | 211
  Male | 130 | 47 | 177
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Germany | 275 | 113 | 388

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity
Description: Sensitivity (true positive rate) of antigen test in symptomatic participants compared with reference standard PCR test (at a threshold of >=10^6 RNA copies/ml for positive PCR results)
Time Frame: Through study completion, an average of 1 1/2 month
Population: 8 symptomatic participants with low RNA copy number were excluded for the calculation of the primary endpoint As this endpoint only considers the sensitivity in symptomatic participants, no numbers are shown for the asymptomatic group
Measure: Number (95% Confidence Interval); unit: percentage of true cases
Arm/Group | Symptomatic | Asymptomatic
Number analyzed (Participants) | 264 | 0
percentage of true cases | 96.7 [88.8 to 99.1] |

2. Primary Outcome: Specificity
Description: Specificity (true negative rate) of antigen test in symptomatic participants compared with reference standard PCR test (at a threshold of >=10^6 RNA copies/ml for positive PCR results)
Time Frame: Through study completion, an average of 1 1/2 month
Population: 8 symptomatic participants were excluded due to low RNA copy number As this endpoint only considers the specificity in symptomatic participants, no numbers are shown for the asymptomatic group
Measure: Number (95% Confidence Interval); unit: percentage of true negative cases
Arm/Group | Symptomatic | Asymptomatic
Number analyzed (Participants) | 264 | 0
percentage of true negative cases | 99.5 [97.3 to 99.9] |

3. Secondary Outcome: Sensitivity in Relation to the Cycle Threshold Value of the Reference RT-PCR (in the Symptomatic Group)
Description: Description of relationship between cycle threshold value of the reference RT-PCR and Dräger test performance.
  Presented is the sensitivity(true positive rate) in the symptomatic group at a cycle threshold of <22
Time Frame: Through study completion, an average of 1 1/2 month
Population: For the calculation of this endpoint only the PCR-positive participants from the symptomatic group were counted.
Measure: Number (95% Confidence Interval); unit: percentage of true positive cases
Arm/Group | Symptomatic | Asymptomatic
Number analyzed (Participants) | 69 | 0
percentage of true positive cases | 97.8 [88.7 to 99.6] |

4. Secondary Outcome: Sensitivity in Relation to the Time Since Symptom Onset (in the Symptomatic Group)
Description: Description of relationship between days since symptom onset and Dräger test performance.
  Presented is the sensitivity(true positive rate) in the symptomatic group at days since symptom onset <5
Time Frame: Through study completion, an average of 1 1/2 month
Population: For the calculation of this endpoint only the PCR-positive participants from the symptomatic group were counted.
Measure: Number (95% Confidence Interval); unit: percentage of true positive cases
Arm/Group | Symptomatic | Asymptomatic
Number analyzed (Participants) | 69 | 0
percentage of true positive cases | 90.9 [80.4 to 96.1] |

5. Secondary Outcome: Specificity in Asymptomatic Participants
Description: Specificity of the antigen test in at least 100 asymptomatic participants
Time Frame: Through study completion, an average of 1 1/2 month
Population: For the calculation of this endpoint only the PCR-negative participants from the asymptomatic group were counted.
Measure: Number (95% Confidence Interval); unit: percentage of true negative cases
Arm/Group | Symptomatic | Asymptomatic
Number analyzed (Participants) | 0 | 105
percentage of true negative cases |  | 100 [96.5 to 100]

6. Secondary Outcome: Frequency of Nosebleed or Unbearable Pain During or Immediately After Specimen Collection
Description: Record of occurrence of lasting nosebleed or unbearable pain during or immediately after specimen collection
Time Frame: Through study completion, an average of 1 1/2 month
Measure: Count of Participants; unit: Participants
Arm/Group | Symptomatic | Asymptomatic
Number analyzed (Participants) | 275 | 113
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Symptomatic | Asymptomatic
All-Cause Mortality (participants affected / at risk) | 0/275 | 0/113
Serious Adverse Events (participants affected / at risk) | 0/275 | 0/113
Other Adverse Events (participants affected / at risk) | 0/275 | 0/113

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-11): https://cdn.clinicaltrials.gov/large-docs/93/NCT04698993/Prot_SAP_001.pdf